CLINICAL TRIAL: NCT04565938
Title: Clinical Performance of a One-step Self-etch Adhesive in Non-carious Cervical Lesions at 2 Years
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Effie Pappa, Dr, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 118/12-3-2009
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Non-carious Cervical Lesions; Adhesive Performance
Keywords: One-step Adhesive; Self-etch Adhesive; Non-carious cervical lesions; Clinical trial
MeSH Terms: interventions — Composite Resins

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- one-step self-etch adhesive with enamel etching (Experimental): Non carious cervical lesions which will receive composite-resin restorations, with one-step self-etch adhesive with enamel etching
  Interventions: Procedure: Application of adhesive for the restoration of dental lesions with resin composite
- one-step self-etch adhesive without enamel etching (Experimental): Non carious cervical lesions which will receive composite-resin restorations, with one-step self-etch adhesive without enamel etching
  Interventions: Procedure: Application of adhesive for the restoration of dental lesions with resin composite
- two-step etch-and-rinse adhesive (Experimental): Non carious cervical lesions which will receive composite-resin restorations, with a two step etch-and-rinse adhesive
  Interventions: Procedure: Application of adhesive for the restoration of dental lesions with resin composite

INTERVENTIONS:
Procedure: Application of adhesive for the restoration of dental lesions with resin composite — 1. Mechanical removal of sclerotic dentin with a round bur
  2. Enamel beveling
  3. Enamel (30sec) and dentin (15sec) etching with phosphoric acid
  4. Application of ExciTE (Ivoclar/Vivadent, AG, Shaan, Lichtenstein) and curing for 10sec with 800mW/cm2 light intensity (Cure TC-01, Spring Health Products, Inc, Norristown, PA, USA)
  5. Composite-resin application using a transparent cervical matrix (Kerr-Hawe, Orange, CA, USA) and curing for 40sec
  6. Finishing and polishing
  Arms: two-step etch-and-rinse adhesive
Procedure: Application of adhesive for the restoration of dental lesions with resin composite — 1. Mechanical removal of sclerotic dentin with a round bur
  2. Enamel beveling
  3. Application of AdheSE One (Ivoclar/Vivadent, AG, Shaan, Lichtenstein) and curing for 10sec
  4. Composite-resin application using a transparent cervical matrix and curing for 40sec
  5. Finishing and polishing
  Arms: one-step self-etch adhesive without enamel etching
Procedure: Application of adhesive for the restoration of dental lesions with resin composite — 1. Mechanical removal of sclerotic dentin with a round bur
  2. Enamel beveling
  3. Enamel (30sec) etching with phosphoric acid
  4. Application of AdheSE One and curing for 10sec
  5. Composite-resin application using a transparent cervical matrix and curing for 40sec
  6. Finishing and polishing
  Arms: one-step self-etch adhesive with enamel etching

SUMMARY:
Objectives: One-step self-etch adhesives are the latest adhesives introduced into the market. The aim of this randomized controlled clinical trial was to test the hypothesis that a one-step self-etch adhesive performs equally well as a two-step etch-and-rinse adhesive.

Materials and methods: Thirty two patients with 96 non-carious cervical lesions received composite-resin restorations (Tetric Evo Ceram - Ivoclar/Vivadent), which were bonded either with a one-step self-etch adhesive (AdheSE One - Ivoclar/Vivadent) with or without enamel etching, or with a two-step etch-and-rinse adhesive (ExiTE - Ivoclar/Vivadent). All restorations were evaluated by two examiners at baseline, 6, 12, 18 and 24 months regarding retention, caries recurrence, marginal integrity and discoloration. Retention loss, severe marginal defects and/or discoloration that needed intervention (repair or replacement) and occurrence of caries, were considered as clinical failures. A logistic regression analysis with generalized estimating equations was used to account for the clustered data (three restorations per patient).

DETAILED DESCRIPTION:
Sample selection Patients, receiving dental treatment in the Clinic of Restorative Dentistry, constituted the selection pool. Written informed consent was obtained from all participants before starting treatment. A total of 32 participants were examined to check if they met the inclusion and exclusion criteria by two precalibrated operative dentistry residents. The qualified patients were recruited in the order in which they reported for the screening session, thus forming a convenience sample.

Patients, irrespective of age and gender, should have at least three non-carious cervical lesions on incisors, canines and premolars of the upper or lower jaw. Each lesion should be located at the cervical third of the buccal side of the tooth, be either at the same level or above the gums, have its cervical wall on dentin, not extend on adjacent surfaces and not exceed 5mm in length, 3mm in height and 1.5mm in depth.

Patients receiving periodontal therapy, presenting high caries activity or TMJ problems needing treatment with mouthguards, were excluded from the study.

A total of thirty two patients with ninety six lesions, were eventually included in the study.

Restoration process

All restorations were performed by only one experienced dentist. All three lesions per patient were restored with Tetric EvoCeram (Ivoclar/Vivadent, AG, Shaan, Lichtenstein) (Table X) following one of next adhesive procedures for each tooth, in a statistical random order:

1. st method 1. Mechanical removal of sclerotic dentin with a round bur 2. Enamel beveling 3. Enamel (30sec) and dentin (15sec) etching with phosphoric acid 4. Application of ExciTE (Ivoclar/Vivadent, AG, Shaan, Lichtenstein) (Table X) and curing for 10sec with 800mW/cm2 light intensity (Cure TC-01, Spring Health Products, Inc, Norristown, PA, USA) 5. Composite-resin application using a transparent cervical matrix (Kerr-Hawe, Orange, CA, USA) and curing for 40sec 6. Finishing and polishing
2. nd method 1. Mechanical removal of sclerotic dentin with a round bur 2. Enamel beveling 3. Application of AdheSE One (Ivoclar/Vivadent, AG, Shaan, Lichtenstein) (Table X) and curing for 10sec 4. Composite-resin application using a transparent cervical matrix and curing for 40sec 5. Finishing and polishing
3. rd method 1. Mechanical removal of sclerotic dentin with a round bur 2. Enamel beveling 3. Enamel (30sec) etching with phosphoric acid 4. Application of AdheSE One and curing for 10sec 5. Composite-resin application using a transparent cervical matrix and curing for 40sec 6. Finishing and polishing

Randomization

The methods were applied in random order (using randomization tables), by which the first randomly selected method was used to restore the tooth with the lowest tooth number (according to the FDI system), the second method was used for the tooth with the second lowest tooth number and the third one for the lowest. In case of more than three lesions, an equal number of restorations with each method was ensured. In instances of an uneven number of restorations placed in one patient, the inequality of number of teeth restored with each method was adjusted for by restoring the lesions with the respective methods in the next patient (again according to the respective randomization tables).

Restoration evaluation

Two experienced and calibrated dentists, not involved with the placement of the restorations and therefore blinded to the group assignment, performed the evaluation. For training purposes, the examiners observed 10 photographs that were representative of each score for each criterion. They evaluated 10 to 15 subjects each on 2 consecutive days. These subjects had cervical restorations and they did not participate in this project. An intraexaminer and interexaminer agreement of at least 85% was necessary before the beginning of the evaluation. All restorations were evaluated at baseline, 6, 12, 18 and 24 months according to ….. criteria. The parameters evaluated were retention of the restoration, marginal integrity, marginal discoloration and recurrent caries (Table X).

The parameters were evaluated using the criteria introduced by Hickel et al. 2007, 2010. The overall clinical effectiveness of the tested adhesives was recorded in terms of retention, marginal integrity, marginal discoloration, caries recurrence. Retention loss, occurrence of caries along the restoration margins, severe marginal defects and/or discoloration that needed clinical intervention (repair or replacement) were considered as clinical failure. The clinical effectiveness of the three methods was compared for the abovementioned parameters.

ELIGIBILITY:
Inclusion Criteria:

At least three non-carious cervical lesions on incisors, canines and premolars of the upper or lower jaw. Each lesion should be located at the cervical third of the buccal side of the tooth, be either at the same level or above the gums, have its cervical wall on dentin, not extend on adjacent surfaces and not exceed 5mm in length, 3mm in height and 1.5mm in depth

Exclusion Criteria:

Patients receiving periodontal therapy, presenting high caries activity or TMJ problems needing treatment with mouthguards, were excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-10 (Estimated)

PRIMARY OUTCOMES:
Retention of the restorations | 2 years
  percentage of retained restorations
Recurrent caries during examination | 2 years
  percentage of lesion with recurrent caries
Marginal adaptation of the restorations | 2 years
  Measured in μm
Marginal discolouration of the restorations | 2 years
  percentage of stained lesions

CONTACTS AND LOCATIONS:
Overall Officials: Effie Pappa, DDs, MSc, PhD, Principal Investigator — University of Athens
Locations (1):
- University of Athenss, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No